CLINICAL TRIAL: NCT00189085
Title: The Effects of Ezetimibe on Postprandial Hyperlipidemia and Endothelial Dysfunction in Patients With the Metabolic Syndrome.
Brief Title: Effects of Ezetimibe on Postprandial Hyperlipidemia and Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EZET
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2004-08

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Ezetimibe, Simvastatin Drug Combination

INTERVENTIONS:
Drug: simvastatin and ezetimibe

SUMMARY:
In the present study the investigators are researching the effects of the cholesterol absorption inhibitor ezetimibe on postprandial lipemia and postprandial endothelial function in patients with the metabolic syndrome. The lipid-lowering effect of high-dose statin monotherapy on fasting lipids is equal to the combination therapy of low-dose statin and ezetimibe.

DETAILED DESCRIPTION:
In patients at high risk for future cardiovascular events, more intensive LDL cholesterol lowering with high doses statin therapy provides greater protection against death or major cardiovascular events than does a standard regimen. Intensive LDL cholesterol lowering can be achieved by high dose statin treatment or with combination therapy of lower doses statin and ezetimibe. However, it is unclear whether this combination therapy results in the same or more beneficial effects on cardiovascular prognosis.

The metabolic syndrome is a cluster of several vascular risk factors (as abdominal obesity, high blood pressure, hypertriglyceridemia, low HDL cholesterol and high fasting glucose). The underlying pathophysiology is still not fully clarified, but insulin resistance seems to be a main characteristic of this syndrome. Subjects with the metabolic syndrome are at increased risk for the development of cardiovascular morbidity and mortality and type II diabetes. The prevalence of the metabolic syndrome is high in patients with clinical manifestations of vascular diseases and is associated with more vascular damage in these patients.

Insulin resistance is linked to endothelial dysfunction and decreased nitric oxide bioavailability by several mechanisms including, inflammation (as reflected by elevated high sensitive C Reactive Protein (hs-CRP) plasma levels), disruption of insulin receptor signalling cascades, increased production of cytokines and activation of the renin angiotensin system. However, other studies do not support an association between insulin resistance and endothelial function, so this mechanism seems controversial.

In the postprandial state, insulin resistance is associated with hyperlipidemia. Postprandial hyperlipidemia may be an important determinant of endothelial dysfunction as well. Remnants of chylomicron and very low density lipoprotein metabolism impair endothelial dependent vasodilatation. In line with the hypothesis that endothelial function can be used as a surrogate endpoint for cardiovascular morbidity, therapeutic modulation of (postprandial) endothelial function may potentially contribute to prevention of cardiovascular disease in patients with the metabolic syndrome.

Statin therapy modulates (postprandial) endothelial function but it is not known whether this is an indirect effect of lipid-lowering or a direct vascular effect of statins influencing the stability and bioavailability of NOS.

AIMS In the present study we propose to investigate the effects of the cholesterol absorption inhibitor ezetimibe on postprandial lipemia and (postprandial) endothelial function in patients with the metabolic syndrome. High-dose statin monotherapy has the same lipid-lowering effect (on fasting lipids) as the combination therapy of low dose statin and ezetimibe. The latter may reduce postprandial lipemia more effectively and may therefore have beneficial effects on postprandial endothelial dysfunction.

Ezetimibe is unlikely to have a direct vascular effect and therefore any observed change in vascular function is due to a change in postprandial lipemia. As secondary objective of the study, this enables us to differentiate between direct and indirect effects of statin therapy on postprandial endothelial function comparing modulation of postprandial endothelial function by monotherapy simvastatin with combination therapy of simvastatin and ezetimibe.

Hypothesis With comparable reduction in fasting plasma lipids, combination therapy of low-dose statin and ezetimibe reduces postprandial lipemia better than high-dose statin monotherapy. This leads to better postprandial endothelial function in patients with the metabolic syndrome.

Objectives

1. To determine the effects of combination therapy of low-dose statin and ezetimibe on postprandial hyperlipidemia compared to high-dose statin monotherapy.
2. To determine the effects of combination therapy of low-dose statin and ezetimibe on postprandial endothelial (dys-)function compared to high-dose statin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female (postmenopausal) patients, 18-70 years of age
2. Diagnosis of the metabolic syndrome according to ATP III criteria(4), including 3 or more of the following metabolic abnormalities:

   * abdominal obesity (waist circumference > 102 cm in men and > 88 cm in women)
   * elevated blood pressure (³ 130 mmHg systolic or ³ 85 mmHg diastolic)
   * hypertriglyceridemia (serum triglycerides ³ 1.70 mmol/L
   * low high-density lipoprotein (HDL) cholesterol (serum HDL-cholesterol <1.04 mmol/L in men and < 1.29 mmol/L in women)
   * high fasting glucose (fasting serum glucose ³ 6.1 mmol/L)
3. Written informed consent

Exclusion Criteria:

1. Smoking
2. Thyroid disease (TSH > 5 mU/L with clinical symptoms of hypothyroidism)
3. Hepatic disease (ASAT or ALAT > 2 times the upper limit of normal)
4. Renal disease (serum creatinine > 1.7 times the upper limit of normal).
5. A history of coronary heart disease, cerebrovascular disease or peripheral arterial disease.
6. Use of lipid lowering therapy
7. Systolic blood pressure ≥ 180 mmHg and /or diastolic blood pressure ≥ 110 mmHg
8. BMI > 35
9. HbA1c > 6.5%
10. Triglycerides > 8.0 mmol/L

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-12; Study Completion 2005-07

PRIMARY OUTCOMES:
Postprandial lipemia | 0, 1, 2 and 4 hours after eating
Postprandial endothelial function | 0 and 4 hours after the meal

CONTACTS AND LOCATIONS:
Overall Officials: Frank LJ Visseren, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- Department of Vascular Medicine UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Westerweel PE, Visseren FL, Hajer GR, Olijhoek JK, Hoefer IE, de Bree P, Rafii S, Doevendans PA, Verhaar MC. Endothelial progenitor cell levels in obese men with the metabolic syndrome and the effect of simvastatin monotherapy vs. simvastatin/ezetimibe combination therapy. Eur Heart J. 2008 Nov;29(22):2808-17. doi: 10.1093/eurheartj/ehn431. Epub 2008 Sep 28. PMID 18824462
- [Derived] Olijhoek JK, Hajer GR, van der Graaf Y, Dallinga-Thie GM, Visseren FL. The effects of low-dose simvastatin and ezetimibe compared to high-dose simvastatin alone on post-fat load endothelial function in patients with metabolic syndrome: a randomized double-blind crossover trial. J Cardiovasc Pharmacol. 2008 Aug;52(2):145-50. doi: 10.1097/FJC.0b013e31817ffe76. PMID 18670365
- [Derived] Hajer GR, Dallinga-Thie GM, van Vark-van der Zee LC, Olijhoek JK, Visseren FL. Lipid-lowering therapy does not affect the postprandial drop in high density lipoprotein-cholesterol (HDL-c) plasma levels in obese men with metabolic syndrome: a randomized double blind crossover trial. Clin Endocrinol (Oxf). 2008 Dec;69(6):870-7. doi: 10.1111/j.1365-2265.2008.03250.x. Epub 2008 Apr 3. PMID 18394022